CLINICAL TRIAL: NCT00240552
Title: An Open-label Phase III Study to Provide Access to Fosamprenavir and to Assess the Long Term Safety and Tolerability of Fosamprenavir Containing Regimens in HIV Infected Patients With Limited Treatment Options
Brief Title: Fosamprenavir Expanded Access
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: APV40005
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: protease inhibitor; Treatment Experienced; amprenavir; fosamprenavir; GW433908; HIV; pro drug
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fosamprenavir

INTERVENTIONS:
Drug: fosamprenavir
Drug: Telzir®
  Other Names: fosamprenavir

SUMMARY:
This open-label study will enable HIV-infected adults with limited treatment options to receive fosamprenavir until commercial supplies are available in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected subjects.
* Subjects must belong to one of the following populations:

  1. Subjects with limited treatment options due to viral resistance, interactions, or tolerability issues with other antiretroviral drugs.
  2. Subjects who already receive amprenavir (Agenerase®)
  3. Subjects for whom once daily dosing of antiretroviral therapy is indicated, including, once daily dosing with fosamprenavir/ritonavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2003-07; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (10):
- Switzerland (10):
  - GSK Investigational Site, Aarau
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Bruderholz
  - GSK Investigational Site, La Chaux-de-Fonds
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Lucerne
  - GSK Investigational Site, Lugano
  - GSK Investigational Site, Sankt Gallen
  - GSK Investigational Site, Zurich